CLINICAL TRIAL: NCT04022863
Title: Early Detection of Ovarian Cancer and Treatment Response by Tumor Educated Platelets (TEP's) and Circulating Tumor DNA (ctDNA)
Brief Title: Ovarium Cancer Detection by TEP's and ctDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gynaecologisch Oncologisch Centrum Zuid (Other)
Collaborators: Leiden University Medical Center (Other); The Netherlands Cancer Institute (Other); Catharina Ziekenhuis Eindhoven (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Jurgen M.J. Piek, principal investigator, Gynaecologisch Oncologisch Centrum Zuid
Other Study IDs: NL68037.100.18
Record Dates: First submitted 2019-07-09; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Neoplasms
Keywords: TEP; ctDNA; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Tumor educated platelets circulating tumor DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ovarian tumor benign: all pathological proven benign ovarian tumors
  Interventions: Diagnostic Test: TEP; Diagnostic Test: ctDNA
- ovarian tumor borderline: all pathological proven borderline ovarian tumors
  Interventions: Diagnostic Test: TEP; Diagnostic Test: ctDNA
- ovarian tumor malignant: all pathological proven malignant ovarian tumors
  Interventions: Diagnostic Test: TEP; Diagnostic Test: ctDNA

INTERVENTIONS:
Diagnostic Test: TEP — Tumor Educated Platelets
Diagnostic Test: ctDNA — circulating tumor DNA

SUMMARY:
Rationale: Cancer is primarily diagnosed by clinical presentation, imaging and pathological analysis of tissue biopsies, increasingly supported by molecular diagnostics tests. However, late diagnosis and misdiagnosis due to limitations of tissue biopsy acquisition remains a major problem. Therefore, a general blood test to pinpoint cancer early and adequately can be considered the 'Holy Grail', because diagnosis in an earlier stage significantly improves the chance of cure from cancer. Several blood-based sources are currently being evaluated as liquid biopsies, including circulating tumor (ct) DNA and circulating tumor cells, but none of these have been implemented for primary (multiclass) cancer diagnostics. Protein tumor markers have been used for decades in diagnosis and monitoring of treatment response in different cancers. Tumor-educated platelets (TEPs) can function as potential blood-based source for (early) cancer diagnostics. Blood platelets are implicated in hemostasis and wound healing. Platelets have recently emerged as central players and immediate responders in the systemic and local responses to tumor growth. Confrontation of platelets by tumor cells via transfer of tumor-associated molecules ('education') results in the sequestration of these molecules (derived from both tumor and its micro-environment), causing a distinct platelet messenger Ribonucleic acid (mRNA) profile. We have previously shown that platelets acquire glioblastoma and prostate cancer mRNA biomarkers and that glioblastoma TEP mRNA profiles harbour diagnostic potential. Furthermore, circulating tumor desoxyrubonucleic acid (ctDNA) has recently been implicated as biomarker for therapy effectiveness and survival. Objective: develop and evaluate the potential of combination of tumor markers, TEPs and ctDNA as liquid biomarkers for (early) ovarium cancer diagnostics and as markers for therapy response and survival. Study design: investigator-initiated, longitudinal, observational study. Study population: patients suspected of having ovarium cancer and are therefore planned for surgery. Main study parameters/endpoints: The difference in biomarker profile from benign ovarium lesions versus cancerous lesions. Nature and extent of the burden and risks associated with participation, benefit and group relatedness. There is no extra burden/risk for the patients in this study. Three extra vials of blood.

DETAILED DESCRIPTION:
Cancer is primarily diagnosed by clinical presentation, radiology, biochemical tests and pathological analysis of tumor tissue, increasingly supported by molecular diagnostic tests. Molecular profiling of tumor tissue samples has emerged as a potential cancer classifying method. In order to overcome limitations of tissue acquisition the use of blood-based liquid biopsies has been suggested. Several blood-based sources are currently being evaluated as liquid biopsies, including plasma DNA and circulating tumor cells. So far, implementation of liquid biopsies for early detection of cancer has been hampered by non-specificity of these sources to pinpoint the nature of the primary tumor. It has been reported that tumor-educated platelets (TEPs) may enable blood-based cancer diagnostics. Platelets are circulating anucleated cell fragments that originate from megakaryocytes in bone marrow, and are traditionally known for their role in hemostasis and initiation of wound healing. More recently, platelets have emerged as central players in the systemic and local responses to tumor growth. Confrontation of platelets with tumor cells via transfer of tumor-associated biomolecules ('education') is an emerging concept and results in the sequestration of such biomolecules. Moreover, external stimuli, such as activation of platelet surface receptors and lipopolysaccharide-mediated platelet activation induce specific splicing of pre-mRNAs in circulating platelets. Platelets may also undergo queue-specific splice events in response to signals released by cancer cells and the tumor microenvironment -such as stromal and immune cells-. The combination of specific splice events in response to external signals and the capacity of platelets to directly ingest (spliced) circulating mRNA can provide TEPs with a highly dynamic mRNA repertoire, with potential applicability to cancer diagnostics. Additionally, the value of other biomarkers that can be derived from a liquid biopsy will be tested in this study. In addition, recently a hallmark paper has shown that combinations of protein tumor markers and ctDNA analysis could discriminate persons with different types of cancer from healthy controls with on average 70% sensitivity (at 99% specificity). In the case of ovarium cancer the sensitivity was 98%. Obvious advantages of liquid biopsy compared to tissue biopsy is the easy accessibility of the material to be obtained and the fact that tumor derived material in blood may cover the cancer heterogeneity where a tissue biopsy is limited to the alterations in the tumor punctured. Therefore, this study investigates the clinical value of longitudinal assessment of liquid biopsy-derived information in diagnosis and monitoring of treatment response in patients suspected of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of ovarian cancer.

Exclusion Criteria:

* Previous intraabdominal malignancies in the history

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with ovarian tumors
Study Population: all women presenting with an ovarian tumor of unknown nature
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of TEP's to determine the nature of an ovarian tumor | 1 month
  Prior to operation blood will be drawn of patients with an ovarian tumor. TEP's will be analysed as described before.
accuracy of ctDNA to determine the nature of an ovarian tumor | 1 month
  Prior to operation blood will be drawn of patients with an ovarian tumor. CtDNA will be analysed as described before.
accuracy of ctDNA to predict treatment response in ovarian cancer | 1 month
  Prior to debulking operation and pre and post chemotherapy ctDNA will be analysed in blood from patients with ovarian cancer as described before.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wurdinger, PhD, Principal Investigator — Amsterdam UMC loc VUmc
Locations (3):
- Netherlands (3):
  - Catharina hospital, Eindhoven, North Brabant
  - Netherlands Cancer Institute, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, North Holland

IPD SHARING:
Plan to Share IPD: Undecided